CLINICAL TRIAL: NCT04355546
Title: A Prospective Non-interventional Trial on COPD Patients' Health Related Quality of Life Under a Fixed LAMA/LABA/ICS Triple Therapy and Characterization of Determinants of Treatment Adherence
Brief Title: Non-interventional Study Related to Fixed LAMA/LABA/ICS Triple Therapy
Acronym: TriOptimize
Status: Completed | Type: Observational
Sponsor: Chiesi UK (Industry)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NIS 004 Pn
Record Dates: First submitted 2020-04-20; First posted 2020-04-21 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: Trimbow 87/5/9 pMDI for COPD prescribed according to licensed indication
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — As this is a Non-interventional trial, only data obtained within the current routine management of COPD at outpatient respiratory centres or GP centres will be documented.

SUMMARY:
This is a prospective non-interventional trial to measure the health related quality of life of patients with chronic obstructive pulmonary disease (COPD) on a fixed LAMA/LABA/ICS triple therapy (Trimbow®) and characterisation of determinants of treatment adherence.

DETAILED DESCRIPTION:
The primary goal of COPD therapy is the prevention of exacerbations and clinical deterioration. To achieve these goals, treatment adherence (i.e. taking medication as prescribed) is important. However, non-adherence (not taking medication as prescribed) is common in COPD and can be affected by lifestyle changes or use of multiple inhalers.

The effects of Trimbow® on patients' health related quality of life, adherence and clinical outcomes have not been assessed in a UK real-world setting. This non-interventional trial aims to collect data from COPD patients under routine care over a 6 month period, for whom their doctors has decided to prescribe Trimbow® as per the authorised indication. We plan to investigate any changes in quality of life, as well as changes in lung function and the need for any additional therapy over 6 months. We also plan to investigate the adherence or reasons for non-adherence to Trimbow® as used in everyday routine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe COPD (with and without concomitant asthma)
2. Physician decision to start therapy with Trimbow as per its current marketing authorisation; the treatment decision should be made independently from participation in this Non-Interventional Trial
3. Patients with at least one COPD exacerbation within the previous 12 months
4. Patients willing and able to sign informed consent for use of their pseudonymised clinical data within the present Non-Interventional Trial

Exclusion Criteria:

1. Patients hospitalised due to an exacerbation of their COPD within the last 4 weeks prior to enrolment
2. Participation within an interventional clinical trial within 30 days prior to enrolment into the present Non-Interventional Trial

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will only be included in the Non-Interventional Trial if Trimbow® has been prescribed in line with its current marketing authorisation and the guidance specified in the summary of product characteristics (SmPC).
  Physicians are urged to offer enrolment to all of their eligible patients consecutively as they present for their routine visit, and not select patients from their patient database.
  Eligible patients may only be included in the NIT after providing written (witnessed, where required by law or regulation), IEC-approved informed consent, or, if incapable of doing so, after such consent has been provided by a legally acceptable representative of the patient.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Assess change in health related quality of life in COPD patients prescribed Trimbow | 6 months
  Change in total CAT score between baseline and after 6 months of treatment.

SECONDARY OUTCOMES:
Assess adherence to COPD therapy | 6 months
  changes in adherence scores (assessed by means of TAI questionnaire),
changes in relevant spirometry parameters | 6 months
  between baseline, e.g. FEV1, FVC
incidence of clinical events | 6 months
  e.g. exacerbations
Compare requirement of rescue medication and alteration of COPD therapy | 6 months
  incidence of COPD medication changes and rescue medication use medication changes and rescue medication use

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Heart and Chest Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No